CLINICAL TRIAL: NCT05834218
Title: Comparative Effects of Split-body and Full-body Resistance Training on Strength and Functional Performance in Amateur Cricket Players
Brief Title: Comparing Split-Body and Full-Body Resistance Training in Amateur Cricket Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0410
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Sports Physical Therapy
Keywords: Resistance training, cricket, Strength

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- split-body resistance training (Experimental): Split-group training regime:
  Day 1 (Leg press, Stiffed-legged deadlift, Leg extension, Hip thrust) 3x12 repetitions for each exercise Day 2 ( Lat pulldown, Bench press, Cabled seated row)3x12 reps (Triceps press and biceps curls in cable (superset) Day 3 (Day 1 exercise repeated) Day 4 (Day 2 exercise repeated)
  Interventions: Other: split body resistance training
- Full body resistance training (Active Comparator): Full body training regime:
  Day 1 (Leg press, Stiffed-legged deadlift, Leg extension, Hip thrust, Lat pulldown, Bench press, Cabled seated) 3x12 reps for each exercise, (Triceps press and biceps curls in cable (superset) Day 2 (Repeat first day exercise)
  Interventions: Other: full body resistance training

INTERVENTIONS:
Other: split body resistance training — Split-group training regime:
  Day 1 (Leg press, Stiffed-legged deadlift, Leg extension, Hip thrust) 3x12 repetitions for each exercise Day 2 ( Lat pulldown, Bench press, Cabled seated row)3x12 reps (Triceps press and biceps curls in cable (superset) Day 3 (Day 1 exercise repeated) Day 4 (Day 2 exercise repeated)
  Arms: split-body resistance training
Other: full body resistance training — Full body training regime:
  Day 1 (Leg press, Stiffed-legged deadlift, Leg extension, Hip thrust, Lat pulldown, Bench press, Cabled seated) 3x12 reps for each exercise, (Triceps press and biceps curls in cable (superset) Day 2 (Repeat first day exercise)
  Arms: Full body resistance training

SUMMARY:
Cricket is an extremely demanding sport. At an elite level, players are often required to perform at their limits of speed, agility, flexibility, endurance and strength. On top of all of this, players must maintain a high state of concentration in order to meet the tactical/mental demands of dealing with their opponents. In young cricket players, the most important attributes are high levels of skill. A long-term commitment to endurance and strength training is necessary to reach and maintain a player's full physical potential. The two primary objectives of the resistance program are to prevent injury and enhance the game's abilities. Strength plays a key role in all motor abilities, technical skills and tactical actions. Endurance performance capacity has long been recognized as an important prerequisite for on-field performance for Cricket players.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial in which 28 sample sizes will be taken. The participants will be allocated into two groups of 14 participants in each group. One group will perform split body exercises in which 4 days of training will include and every day a single muscle group will be targeted for example on day one the arm muscles bicep and triceps are included and on day two leg press will include and so on. In the second group whole body resistance exercises will perform in two days for example on day one bench press leg press and other resistance training exercises will be performed. Training will give to both groups for 6 weeks. After 6 weeks we compare both groups by FMS and the Leg press bench press test will perform. Data will be analyzed by using SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* Only male cricketers will be recruited to the study.
* We have to select those individuals which are of ages 20 to 30 years.
* only those individuals will be recruited with no history of any systemic disease.

Exclusion Criteria:

* cricketers who have received surgery in the three years prior to the study or undergone rehabilitation within the past year.
* cricketers who would not commit to full participation in the study's training regimes.
* cricketers who will have any systemic disease which can hinder the training.
* Cricketers currently engaged in strength training as this may confound the study.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-10-22 (Estimated)

PRIMARY OUTCOMES:
Bench Press Test | 6 weeks
  The 1RM test is considered a valid assessment of maximal bench press strength and requires the lifter to push a maximally loaded barbell off their chest from a pause to a fully extended elbow position at approximately eyebrow level
Leg Press Test | 6 weeks
  This test requires the athlete to complete as many leg presses as possible with no rest. The assistant weighs and records the athlete's weight. The athlete warms up for 10 minutes. The assistant loads the barbell with a weight close to the athlete's one repetition maximum load
30 Second Sit to Stand Test | 6 weeks
  Often provides a better picture of the relationship between strength and disability. As the patient does various maneuvers,deficiencies are noted and quantified as much as possible. This test measures the number of times an individual can stand from a chair with no assistance in 30 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Amna Shahid, t-DPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Raiwind Campus, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No